CLINICAL TRIAL: NCT03752736
Title: Sun Safety Skills for Elementary School Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Kristin M. Nord, Clinical Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 46831
Record Dates: First submitted 2018-10-16; First posted 2018-11-26 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Sunburn; Skin Cancer Prevention
Keywords: Sunscreen; Sun protection; Education; skin cancer; school-aged children; prevention
MeSH Terms: conditions — Sunburn; Skin Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Extended intervention (Active Comparator): Upon completion of the two-week baseline period and two-week standard intervention period, the two classrooms assigned to the Extended intervention condition will receive the "I wear sunscreen everyday" song-based video intervention daily for two additional weeks.
  Interventions: Behavioral: "I wear sunscreen everyday" song-based video
- Maintenance (No Intervention): The two classrooms assigned to the Maintenance condition will continue to receive a two- minute window for sunscreen application, but no "I wear sunscreen everyday" song-based video instruction.
  Change trajectories from Time 3-Time 4 (two-week follow up) will be compared by follow-up assignment condition and will provide preliminary information about dosing and maintenance effects.

INTERVENTIONS:
Behavioral: "I wear sunscreen everyday" song-based video — All four classes (arms) will be shown (sitting on carpet, not participating) a 2-3 minute song-based video titled "I wear sunscreen everyday" in which they observe elementary age children applying sunscreen in a systematic fashion. Following the viewing, classes will be administered this video guided, song- based intervention while their teacher documents their independent participation using our classroom map data collection sheet.
  Arms: Extended intervention

SUMMARY:
The overarching goal of this work is to pilot-test a song-based instructional video designed to help elementary school (kindergarten) age children independently apply sunscreen effectively (i.e., covers all needed areas), efficiently (i.e., can be accomplished in 2-3 minutes), consistently (i.e., continues to apply sunscreen routinely before recess both during and after the intervention), without impacting classroom function (i.e., no mess). The video is also designed to encourage use of hats and sunglasses. The outcomes of interest include identification of "gaps" in skills that are consistent for this age group (i.e., commonly miss application to the back of neck), areas of learning refinement (i.e., generalization of skills with different outfits on), and flexibility in terms of adapting practice (i.e., can they do it without the video). The investigators hope that this pilot project will pave the way for broader clinical / educational implementation of this intervention within schools.

DETAILED DESCRIPTION:
The investigators will use an unblinded, open label, A-B design with a randomized follow-up period to evaluate the study objectives. The primary aim is to characterize the proportion of students (per class and total, or across classes) who productively engage in the in-classroom sunscreen application tasks when using the video guided sunscreen intervention (i.e., success is defined as any appropriate participation with video guided tasks, completing tasks and putting sunscreen away, sitting down by end of 2 minute, 42 second video intervention) relative to the proportion who achieve success (i.e., any appropriate effort to apply sunscreen, put away sunscreen and sit down within a two minute window) WITHOUT use of the video.

One hundred eight kindergarten students across four kindergarten classrooms (N = 27 per class) will complete a two-week baseline period in which the participants are provide a 2-minute window and allowed access to their sunscreen without instruction. Classroom teachers, trained to score our primary outcome (child does/does not complete this task within two-minute window), will evaluate outcomes for each child daily for two weeks (baseline period). Percentage of students who are able to complete this task is our primary endpoint. Change trajectories from beginning to end of the baseline period (Time 1/Day 1 - Time 2/Day 10) and from the beginning to end of treatment (Time 2 - Time 3) will be calculated for each class. The average percentage of the second week in the baseline period and the second week in the intervention period will be used to calculate the successful rate for each period with 95% confidence intervals.

To address a subsidiary aim, related to whether or not student competence with sunscreen application (systematic, % of body covered / body parts neglected, and completeness of coverage of face) is impacted by the video intervention, a randomly selected subset of students will be evaluated by a trained member of the study team for competence of application at Time 1,2, 3 and 4. Changes trajectories will be calculated by class for this subset of students.

At the study outset, all four classrooms will be randomized to either an "extended intervention" (EI) or "maintenance" (M) condition using a 1:1 randomization scheme. This will offer some descriptive, feasibility data regarding the tolerability of randomization by classroom, and a preliminary look at dose-response trends and short-term maintenance effects. Upon completion of the two-week baseline period and two-week standard intervention period, the two classrooms assigned to the EI condition will receive the video-based intervention for two additional weeks and the two classrooms assigned to the M condition will continue to receive a two- minute window for sunscreen application, but no video-based instruction. Change trajectories from Time 3-Time 4 (two-week follow up) will be compared by follow-up assignment condition and will provide preliminary information about dosing and maintenance effects.

Student, teacher, parent and administrator perceptions of the acceptability, value and utility of the intervention will be assessed at a single time point at the conclusion of the study.

Study Setting and Participants:

General Education Kindergarten students who meet all study eligibility requirements (i.e., including health requirements appropriate to the use of sunscreen) and who assent to participate and who receive parental consent to participate at Sedgwick Elementary School will be included in the present study. Special education students who are mainstreamed may also be considered eligible to participate via consensus from both parent and teacher.

Recruitment and screening: Recruitment efforts will include collaborative (research team + kinder teachers) efforts to provide parents an overview of the study goals and objectives, and to obtain consent/assent. The investigators will plan to have a parent-focused meeting in the weeks prior to the commencement of the study.

Intervention: The song-based video guided sun screen intervention is 2-3 minutes long, with 30 seconds allotted at the beginning for students to prepare their sunscreen materials and get ready, two minutes of instruction that guides their application of sunscreen to all exposed areas of skin starting with their head and working systematically down to their feet, and then 30 seconds of guided instruction for putting the sunscreen materials away and sitting back down at their desks.

ELIGIBILITY:
Inclusion Criteria:

* General education Kinder students (Sedgwick Elementary School in 2018-2019).
* Child assent and parental consent are required to participate.

Exclusion Criteria:

* Non-general education status;
* significant medical, mental health and/or behavioral problem
* child refusal of assent or parental refusal of consent;
* known or identified allergy to ingredients in sunscreen;
* moving out of the grade or school during the intervention or follow-up period;
* participation in a concurrent sunscreen intervention protocol are exclusionary criteria.

Ages: 5 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 96 (Actual)
Dates: Start 2019-02-25 (Actual); Primary Completion 2019-04-11 (Actual); Study Completion 2019-05-23 (Actual)

PRIMARY OUTCOMES:
Teacher Ratings of Kinder Students' Successful/Not Successful Self-Application of Sunscreen. | Baseline to Posttreatment (Time 1 - Time 2; each Time is up to 15 minutes and separated by 2 weeks)
  Change in the proportion of kindergarten students who successfully complete independent self-application of sunscreen within the allotted 2.5 minute time window from baseline (Time 1) to posttreatment (Time 2). Successful completion of the sun screen task (i.e., Kinder Students' self-application of sunscreen within the 2.5 minute window allotted by the intervention) will be determined via direct observation by the classroom teacher. Teachers will be formally trained by the study staff to rate student performance (i.e., successful/not successful) with self-application of sunscreen per a manualized study protocol.

SECONDARY OUTCOMES:
Teacher Identified Barriers to Kinder Student Self-Application of Sunscreen | Baseline to Posttreatment (Time 1 - Time 2; each Time is up to 15 minutes and separated by 2 weeks)
  Teacher identified barriers, or the cognitive, emotional, behavioral, environmental, factors that interfered with a student's successful completion of the self-application of sunscreen task will be recorded by the classroom teacher daily during the sunscreen intervention. This descriptive outcome will be qualitative (i.e., teacher generated list).
Teacher, parent and administrator perceptions of intervention utility. | Posttreatment (Time 2; up to 15 minutes)
  Teacher, parents and administrators respond to a single item question, "In your opinion, how useful was this intervention in terms of getting students engaged in sun protective behavior?" This single item is modeled after utility questions used in health services research and educational research, and will be scored on an 11-point likert type scale, where "0" indicates not at all useful; and "10" indicates very useful.
Teacher, parent and administrator perceptions of intervention value. | Posttreatment (Time 2; up to 15 minutes)
  Teacher, parents and administrators respond to a single item question "In your opinion, how valuable was this intervention to your overall curriculum? This single item is modeled after value questions used in health services and educational research and will be Responses will be scored on an 11-point likert type scale, where a score of "0" indicates not at all valuable and a score of "10" indicates very valuable.
Student perceptions of intervention likability | Posttreatment (Time 2; up to 15 minutes)
  Kinder students respond to a single item question "Did you like the sunscreen video? " As Kinder students are not proficient readers, this question will be read aloud to the class, and students will respond individually by casting a "secret ballot" in a voting booth set up in the classroom- -under the direct supervision of the study staff. "Yes" votes will be cast using a piece of paper with a happy face on it; "no" votes will be cast using a piece of paper with a sad face on it. In this way, students can respond individually to this question without having to read, tell their answer to the teacher, and without undue influence of their peers. Results will be tallied by class.

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Nord, MD, Principal Investigator — Stanford University
Locations (1):
- Sedgwick Elementary School, Cupertino, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee GH, Bae GH, Barnes LA, Pol-Rodriguez MM, Ransohoff KJ, Nord KM, Lu Y, Cannell B, Weitlauf JC. The Sunscreen for Kindergarteners (SKIN) Study trial protocol. Contemp Clin Trials. 2021 Aug;107:106480. doi: 10.1016/j.cct.2021.106480. Epub 2021 Jun 11. PMID 34126263